CLINICAL TRIAL: NCT00847015
Title: Phase II Study of Gemcitabine, Cisplatin, and Sunitinib (GC-S) as Neoadjuvant Chemotherapy in Patients With Muscle-Invasive Bladder Cancer
Brief Title: Gemcitabine, Cisplatin, and Sunitinib (GC-S) as Neoadjuvant Chemotherapy in Patients With Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-159
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Bladder Cancer; Urinary Bladder
Keywords: Bladder; Urinary; CISPLATIN; GEMCITABINE; SU011248 (Sunitinib Malate); 08-159
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Cisplatin, and Sunitinib (Experimental): This is a phase II study of GCS (Gemcitabine, Cisplatin, and Sunitinib) as neoadjuvant chemotherapy in patients with muscle-invasive urothelial carcinoma of the bladder. Patients with muscle invasive urothelial carcinoma who are candidates for radical cystectomy will be enrolled.
  Interventions: Drug: Sunitinib; Drug: Gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: Sunitinib — Sunitinib will be administered at a dose of 25mg orally once daily for 2 consecutive weeks followed by a 1 week rest period.
Drug: Gemcitabine — Gemcitabine 1,000 mg/m^2
Drug: cisplatin — cisplatin 35 mg/m^2 will be administered intravenously on days 1 and 8.

SUMMARY:
The purpose of this study is to find out if using the combination of standard chemotherapy (gemcitabine and cisplatin) plus this new targeted pill (sunitinib) can help shrink your tumor before you undergo surgery for your bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed muscle invasive transitional cell carcinoma of the bladder at MSKCC.
* Clinical stage T2-T4a N0/X M0 disease.
* Medically appropriate candidate for radical cystectomy as per MSKCC attending urologic oncologist.
* Karnofsky Performance Status ≥ 70%.
* Age ≥ 18 years of age.
* Required Initial Laboratory Values:

  * Absolute neutrophil count ≥ 1500 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 9.0g/dL
  * Bilirubin ≤ 1.5 the upper limit of normal (ULN) for the institution
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN for the institution
  * Alkaline phosphatase ≤ 2.5 x ULN for the institution
  * Serum creatinine ≤ 1.5 mg/dL
* Estimated glomerular filtration rate ≥ 60 ml/min/1.73m2 using the CKD-EPI equation:
* eGFR = 141 x min(Scr/k, 1)a x max(Scr/k, 1)-1.209 x 0.993Age
* x 1.018 [if female] x 1.159 [if black]
* Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1.
* If female of childbearing potential, pregnancy test is negative.
* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial.

Exclusion Criteria:

* Prior systemic chemotherapy (prior intravesical therapy is allowed)
* Prior radiation therapy to the bladder
* Evidence of NYHA functional class III or IV heart disease.
* Serious intercurrent medical or psychiatric illness, including serious active infection.
* Preexisting sensory grade 3 neuropathy
* Major surgery or radiation therapy < 4 weeks of starting study treatment.
* Concomitant use of any other investigational drugs
* Any of the following within the 6 months prior to study drug administration:

myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.

* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade ≥ 2.
* Prolonged QTc interval on baseline EKG (>450 msec for males and >470 msec for females).
* Uncontrolled hypertension (>150/100 mmHg despite optimal medical therapy).
* Pre-existing thyroid abnormality, with thyroid function tests that cannot be maintained in the normal range with medication.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Ongoing treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg po daily for thromboembolic prophylaxis is allowed).
* Pregnancy or breast-feeding. Patients must be surgically sterile or be postmenopausal,or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Male patients must be surgically sterile or agree to use effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine, Cisplatin, and Sunitinib: This is a phase II study of GCS (Gemcitabine, Cisplatin, and Sunitinib) as neoadjuvant chemotherapy in patients with muscle-invasive urothelial carcinoma of the bladder. Patients with muscle invasive urothelial carcinoma who are candidates for radical cystectomy will be enrolled.
  Gemcitabine, Cisplatin, and Sunitinib: Patients will receive four cycles of GCS administered every 21 days followed by radical cystectomy. Sunitinib will be administered at a dose of 25mg orally once daily for 2 consecutive weeks followed by a 1 week rest period. Gemcitabine 1,000 mg/m2 and cisplatin 35 mg/m2 will be administered intravenously on days 1 and 8.
Period: Overall Study
Arm/Group | Gemcitabine, Cisplatin, and Sunitinib
Started | 18
Completed | 15
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — declined any surgery | 1
Not completed — partial cystectomy vs radical cystectomy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Cisplatin, and Sunitinib
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: The Pathologic Complete Response Rate (<pT0) of Neoadjuvant GCS Regimen in Patients With Muscle-invasive Bladder Cancer.
Description: Complete pathologic response to neoadjuvant GCS is the primary endpoint is defined as the absence of carcinoma (pT0 disease) and the absence of microscopic lymph node metastases (N0) on the final cystectomy specimen.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine, Cisplatin, and Sunitinib
Number analyzed (Participants) | 15
percentage of participants | 6.67 [.34 to 29.8]

2. Secondary Outcome: The Pathologic Response Rate (<pT2) of Neoadjuvant GCS Regimen in Patients With Muscle-invasive Bladder Cancer.
Description: is defined as the absence of muscle invasive carcinoma (<pT2 disease) and the absence of microscopic lymph node metastases (N0) on the final cystectomy specimen.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine, Cisplatin, and Sunitinib
Number analyzed (Participants) | 15
percentage of participants | 33 [15 to 58]

3. Secondary Outcome: The Time to Disease Progression in Patients With Muscle Invasive Urothelial Carcinoma of the Bladder Treated With Neoadjuvant GCS Followed by Radical Cystectomy.
Description: The time to disease progression is measured from the time of initiation of chemotherapy until the first date that systemic recurrence is objectively documented. Systemic recurrence for this trial is defined as either metastatic or local pelvic recurrence.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Cisplatin, and Sunitinib
Number analyzed (Participants) | 15
months | 10 [3.5 to NA] — This number could not be calculated as three participants are deceased.

ADVERSE EVENTS:
Arm/Group | Gemcitabine, Cisplatin, and Sunitinib
Serious Adverse Events (participants affected / at risk) | 14/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Cisplatin, and Sunitinib (N=18)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Neutrophil count decrease (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Cisplatin, and Sunitinib (N=18)
Anemia (Blood and lymphatic system disorders) | 11 (11)
Neutrophil count decreased (Investigations) | 6 (6)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombotic events (Vascular disorders) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 8 (18)
Leukocytes (total WBC) (Cardiac disorders) | 6 (25)
Lymphopenia (Investigations) | 3 (5)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (3)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6 (34)
Platelets (Investigations) | 6 (16)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes